CLINICAL TRIAL: NCT05977894
Title: Wellbeing Monitoring During Sequential Reduced Environmental Stimulation-Floatation
Brief Title: Floatation Experience in Nurses and Physicians
Status: Enrolling by invitation | Type: Observational
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Principal Investigator, C. Michael Dunham, Research Investigator, Mercy Health Ohio
Other Study IDs: 6120-810-1-01
Record Dates: First submitted 2023-07-12; First posted 2023-08-07 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Burnout, Professional; Negative Affect; Positive Affect; Wellbeing; Burnout; Psychological
Keywords: Floatation; Anxiety; Attention; Awareness; Burnout; Relaxation Therapy; Self-concept; Wellbeing
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nurses and physicians: Nurses (registered, practitioner, and anesthetist) and physicians, employed at St. Elizabeth Youngstown Trauma Center, Mercy Health
  Interventions: Other: Reduced Environmental Stimulation Therapy

INTERVENTIONS:
Other: Reduced Environmental Stimulation Therapy — During floatation-REST (Reduced Environmental Stimulation Therapy), the participant enters a tank that is approximately 5 feet wide, 7 feet long and 5 feet high. The tank is filled with a 10 inch height of water containing enough Epsom salt (magnesium sulfate) to create body buoyancy. The water temperature is 93.5 degrees F, an approximate equivalent for normal skin temperature. Ear plugs are used to mitigate sound and the tank is without light illumination to prevent visual stimulation. The sessions are typically 60 minutes in duration. The individual is "Floating-in Solitude, Darkness, Silence, and Thermal-Neutrality." This experience reduces external sensory nervous system input and creates an extraordinarily deep state of mental and physical relaxation.
  Other Names: Floatation-REST

SUMMARY:
The goal of this observational study is to monitor the floatation experience and continue the program as long as deemed important. The main question it aims to answer is: will inventory wellbeing scores increase according to the number of floatation sessions accrued? Nurses (registered, practitioner, and anesthetist) and physicians, employed at St. Elizabeth Youngstown Trauma Center, Mercy Health, will be welcomed to participate in the floatation experience. Participants will be given an option to complete the Wellbeing Inventory survey prior to each floatation session.

DETAILED DESCRIPTION:
The floatation program is a Mercy Health enterprise sponsored by the Mercy Health Mahoning Valley Foundation.The goal of this study is to monitor the floatation experience and continue the program as long as deemed important. The investigators hypothesize that inventory wellbeing scores will increase according to the number of floatation sessions accrued. Nurses (registered, practitioner, and anesthetist) and physicians, employed at St. Elizabeth Youngstown Trauma Center, Mercy Health, will be welcomed to participate in the optional floatation program in Warren, Ohio at no financial cost to them. They will become aware of floatation options through the Mercy Health Be Well wellness program. Floatation monitoring will include assessments of wellbeing, nonstress, and positive affect scores. Participants will be given an option to complete the Wellbeing Inventory survey prior to each floatation session. This will be a self-reporting anonymous process. The investigator will never know the identity of the participant.

ELIGIBILITY:
Inclusion Criteria:

* Nurses and physicians

Exclusion Criteria:

* Any person that is not a physician or nurse at St. Elizabeth Youngstown Hospital

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses (registered, practitioner, and anesthetist) and physicians, employed at St. Elizabeth Youngstown Trauma Center, Mercy Health
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-28 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Change in the inventory wellbeing score | Through study completion, an average of 1 year
  The sum of the positive affect and nonstress scores (range 11-55)

SECONDARY OUTCOMES:
Change in the nonstress score | Through study completion, an average of 1 year
  The sum of the reverse-scored ratings for the 7 negative affect items (range 7-35)
Change in the positive affect score | Through study completion, an average of 1 year
  The sum of the ratings for the 4 positive affect items (range 4-20)

CONTACTS AND LOCATIONS:
Overall Officials: C. Michael Dunham, MD, Principal Investigator — Mercy Health Ohio
Locations (1):
- St. Elizabeth Youngstown Hospital, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The wellbeing scores will be assessed according to the number of floatation sessions undertaken and described in a manuscript to be submitted to a peer-reviewed PubMed journal.
Supporting Information: Study Protocol, SAP
Time Frame: Estimate that a descriptive manuscript will be developed and likely accepted for publication by December 2024.
Access Criteria: Information will be shared through an open access publication.

REFERENCES:
- [Background] Dyrbye LN, Satele D, Sloan J, Shanafelt TD. Utility of a brief screening tool to identify physicians in distress. J Gen Intern Med. 2013 Mar;28(3):421-7. doi: 10.1007/s11606-012-2252-9. Epub 2012 Nov 6. PMID 23129161
- [Background] Dyrbye LN, West CP, Satele D, Boone S, Tan L, Sloan J, Shanafelt TD. Burnout among U.S. medical students, residents, and early career physicians relative to the general U.S. population. Acad Med. 2014 Mar;89(3):443-51. doi: 10.1097/ACM.0000000000000134. PMID 24448053
- [Background] Brazeau CM, Shanafelt T, Durning SJ, Massie FS, Eacker A, Moutier C, Satele DV, Sloan JA, Dyrbye LN. Distress among matriculating medical students relative to the general population. Acad Med. 2014 Nov;89(11):1520-5. doi: 10.1097/ACM.0000000000000482. PMID 25250752
- [Background] Poghosyan L, Clarke SP, Finlayson M, Aiken LH. Nurse burnout and quality of care: cross-national investigation in six countries. Res Nurs Health. 2010 Aug;33(4):288-98. doi: 10.1002/nur.20383. PMID 20645421
- [Background] Vahey DC, Aiken LH, Sloane DM, Clarke SP, Vargas D. Nurse burnout and patient satisfaction. Med Care. 2004 Feb;42(2 Suppl):II57-66. doi: 10.1097/01.mlr.0000109126.50398.5a. PMID 14734943
- [Background] Chang EM, Bidewell JW, Huntington AD, Daly J, Johnson A, Wilson H, Lambert VA, Lambert CE. A survey of role stress, coping and health in Australian and New Zealand hospital nurses. Int J Nurs Stud. 2007 Nov;44(8):1354-62. doi: 10.1016/j.ijnurstu.2006.06.003. Epub 2006 Aug 9. PMID 16901488
- [Background] Lindqvist R, Smeds Alenius L, Griffiths P, Runesdotter S, Tishelman C. Structural characteristics of hospitals and nurse-reported care quality, work environment, burnout and leaving intentions. J Nurs Manag. 2015 Mar;23(2):263-74. doi: 10.1111/jonm.12123. Epub 2013 Sep 19. PMID 24047463
- [Background] Poncet MC, Toullic P, Papazian L, Kentish-Barnes N, Timsit JF, Pochard F, Chevret S, Schlemmer B, Azoulay E. Burnout syndrome in critical care nursing staff. Am J Respir Crit Care Med. 2007 Apr 1;175(7):698-704. doi: 10.1164/rccm.200606-806OC. Epub 2006 Nov 16. PMID 17110646
- [Background] Embriaco N, Papazian L, Kentish-Barnes N, Pochard F, Azoulay E. Burnout syndrome among critical care healthcare workers. Curr Opin Crit Care. 2007 Oct;13(5):482-8. doi: 10.1097/MCC.0b013e3282efd28a. PMID 17762223
- [Background] Chuang CH, Tseng PC, Lin CY, Lin KH, Chen YY. Burnout in the intensive care unit professionals: A systematic review. Medicine (Baltimore). 2016 Dec;95(50):e5629. doi: 10.1097/MD.0000000000005629. PMID 27977605
- [Background] Mealer ML, Shelton A, Berg B, Rothbaum B, Moss M. Increased prevalence of post-traumatic stress disorder symptoms in critical care nurses. Am J Respir Crit Care Med. 2007 Apr 1;175(7):693-7. doi: 10.1164/rccm.200606-735OC. Epub 2006 Dec 21. PMID 17185650
- [Background] Abdo SA, El-Sallamy RM, El-Sherbiny AA, Kabbash IA. Burnout among physicians and nursing staff working in the emergency hospital of Tanta University, Egypt. East Mediterr Health J. 2016 Mar 15;21(12):906-15. doi: 10.26719/2015.21.12.906. PMID 26996364
- [Background] Alqahtani AM, Awadalla NJ, Alsaleem SA, Alsamghan AS, Alsaleem MA. Burnout Syndrome among Emergency Physicians and Nurses in Abha and Khamis Mushait Cities, Aseer Region, Southwestern Saudi Arabia. ScientificWorldJournal. 2019 Feb 18;2019:4515972. doi: 10.1155/2019/4515972. eCollection 2019. PMID 30906233
- [Background] Hamdan M, Hamra AA. Burnout among workers in emergency Departments in Palestinian hospitals: prevalence and associated factors. BMC Health Serv Res. 2017 Jun 15;17(1):407. doi: 10.1186/s12913-017-2356-3. PMID 28619081
- [Background] Hinderer KA, VonRueden KT, Friedmann E, McQuillan KA, Gilmore R, Kramer B, Murray M. Burnout, compassion fatigue, compassion satisfaction, and secondary traumatic stress in trauma nurses. J Trauma Nurs. 2014 Jul-Aug;21(4):160-9. doi: 10.1097/JTN.0000000000000055. PMID 25023839
- [Background] Munnangi S, Dupiton L, Boutin A, Angus LDG. Burnout, Perceived Stress, and Job Satisfaction Among Trauma Nurses at a Level I Safety-Net Trauma Center. J Trauma Nurs. 2018 Jan/Feb;25(1):4-13. doi: 10.1097/JTN.0000000000000335. PMID 29319643
- [Background] Dunham CM, Burger AL, Hileman BM, Chance EA. Psychometric properties of the St. Elizabeth Youngstown hospital wellbeing inventory and non-burnout inventory for physicians and nurses. BMC Psychol. 2019 Jun 17;7(1):36. doi: 10.1186/s40359-019-0316-x. PMID 31208464
- [Background] Kim HS, Yeom HA. The association between spiritual well-being and burnout in intensive care unit nurses: A descriptive study. Intensive Crit Care Nurs. 2018 Jun;46:92-97. doi: 10.1016/j.iccn.2017.11.005. Epub 2018 Apr 3. PMID 29625870
- [Background] Feinstein JS, Khalsa SS, Yeh H, Al Zoubi O, Arevian AC, Wohlrab C, Pantino MK, Cartmell LJ, Simmons WK, Stein MB, Paulus MP. The Elicitation of Relaxation and Interoceptive Awareness Using Floatation Therapy in Individuals With High Anxiety Sensitivity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):555-562. doi: 10.1016/j.bpsc.2018.02.005. Epub 2018 Mar 9. PMID 29656950
- [Background] Flux MC, Fine TH, Poplin T, Al Zoubi O, Schoenhals WA, Schettler J, Refai HH, Naegele J, Wohlrab C, Yeh HW, Lowry CA, Levine JC, Smith R, Khalsa SS, Feinstein JS. Exploring the acute cardiovascular effects of Floatation-REST. Front Neurosci. 2022 Dec 9;16:995594. doi: 10.3389/fnins.2022.995594. eCollection 2022. PMID 36570829
- [Background] Khalsa SS, Moseman SE, Yeh HW, Upshaw V, Persac B, Breese E, Lapidus RC, Chappelle S, Paulus MP, Feinstein JS. Reduced Environmental Stimulation in Anorexia Nervosa: An Early-Phase Clinical Trial. Front Psychol. 2020 Oct 6;11:567499. doi: 10.3389/fpsyg.2020.567499. eCollection 2020. PMID 33123048
- [Background] Schulz P, Kaspar CH. Neuroendocrine and psychological effects of restricted environmental stimulation technique in a flotation tank. Biol Psychol. 1994 Mar;37(2):161-75. doi: 10.1016/0301-0511(94)90029-9. PMID 8003591
- [Background] Caldwell LK, Kraemer WJ, Post EM, Volek JS, Focht BC, Newton RU, Hakkinen K, Maresh CM. Acute Floatation-REST Improves Perceived Recovery After a High-Intensity Resistance Exercise Stress in Trained Men. Med Sci Sports Exerc. 2022 Aug 1;54(8):1371-1381. doi: 10.1249/MSS.0000000000002906. Epub 2022 Apr 6. PMID 35389942
- [Background] Kjellgren A, Sundequist U, Norlander T, Archer T. Effects of flotation-REST on muscle tension pain. Pain Res Manag. 2001 Winter;6(4):181-9. doi: 10.1155/2001/768501. PMID 11854763
- [Background] Kjellgren A, Westman J. Beneficial effects of treatment with sensory isolation in flotation-tank as a preventive health-care intervention - a randomized controlled pilot trial. BMC Complement Altern Med. 2014 Oct 25;14:417. doi: 10.1186/1472-6882-14-417. PMID 25344737
- [Background] Feinstein JS, Khalsa SS, Yeh HW, Wohlrab C, Simmons WK, Stein MB, Paulus MP. Examining the short-term anxiolytic and antidepressant effect of Floatation-REST. PLoS One. 2018 Feb 2;13(2):e0190292. doi: 10.1371/journal.pone.0190292. eCollection 2018. PMID 29394251
- [Background] Jonsson K, Kjellgren A. Promising effects of treatment with flotation-REST (restricted environmental stimulation technique) as an intervention for generalized anxiety disorder (GAD): a randomized controlled pilot trial. BMC Complement Altern Med. 2016 Mar 25;16:108. doi: 10.1186/s12906-016-1089-x. PMID 27016217